CLINICAL TRIAL: NCT00096941
Title: An Open-Label, Multicenter Extension Study of Pertuzumab (rhuMAb 2C4) in Subjects Treated With Pertuzumab in a Previous Genentech-Sponsored Phase II Cancer Study
Brief Title: A Study to Evaluate Subjects Treated With rhuMab 2C4 (Pertuzumab) in a Previous Genentech Phase II Cancer Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOC2664g
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-05

CONDITIONS: Solid Cancers
Keywords: Advanced solid cancers; HER2; EGFR
MeSH Terms: interventions — pertuzumab

ARMS (1):
- Pertuzumab (Experimental): Participants received the same dose of pertuzumab that they received in their parent Phase II trial, either 420 mg or 1050 mg, intravenously on Day 1 of every 3 week cycle until disease progression.
  Interventions: Drug: Pertuzumab

INTERVENTIONS:
Drug: Pertuzumab — Pertuzumab was supplied as a single-use liquid formulation.

SUMMARY:
This is a multicenter, open label extension study. Subjects who have completed treatment in the parent study of pertuzumab, either alone or with a combination agent, and who received at least one dose of pertuzumab in the parent study are eligible for inclusion in this trial if they are continuing to receive clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* ECOG performance status of 0, 1, or 2
* Completion of treatment in a previous Genentech sponsored, Phase II cancer study with pertuzumab, either alone or with a combination agent, in which at least one dose of pertuzumab was received in the parent study
* Less than 3 months since last dose of pertuzumab on the parent study
* Use of an effective means of contraception for men or for women of childbearing potential
* Granulocyte count >= 1500/uL
* Platelet count >= 75,000/uL
* Hemoglobin >= 9 g/dL (hemoglobin may be supported by transfusion or erythropoietin or other approved hematopoietic growth factors; darbepoetin [Aranesp(R)] is permitted)
* Serum bilirubin less than or equal to the upper limit of normal (ULN) (unless due to Gilbert's disease)
* Alkaline phosphatase, AST, and ALT <= 2.5x ULN (<= 5x ULN for subjects with liver metastases; no alkaline phosphatase upper limit for subjects with bone metastases)
* Serum creatinine <= 1.5x ULN
* International normalized ratio (INR) < 1.5 and activated partial thromboplastin time (aPTT) < 1.5x ULN (except for subjects receiving warfarin)

Exclusion Criteria:

* Recent (within the last 3 months), current, or planned participation in a experimental drug study other than a Genentech-sponsored pertuzumab cancer study
* Any unresolved or irreversible NCI-CTC Grade 3 or 4 adverse event or clinically meaningful cardiac adverse event (any grade) that is pertuzumab-related and ongoing from the parent study
* Recent (within the last 3 months) or current treatment with HER pathway inhibitors other than pertuzumab (e.g., Herceptin(R) [Trastuzumab], Iressa<TM> [gefitinib], Tarceva<TM> [erlotinib hydrochloride], C225, CI1033, or TAK165) or other monoclonal antibodies
* Clinical evidence of central nervous system or brain metastases
* Ejection fraction ≤50%, as determined by ECHO (or MUGA)
* Uncontrolled hypercalcemia (> 11.5 mg/dL)
* Recent anthracycline exposure (within the last 3 months) or cumulative exposure of > 360 mg/m^2 doxorubicin or equivalent (i.e., liposomal doxorubicin, > 120 mg/m^2 mitoxantrone, or > 90 mg/m^2 idarubicin)
* Ongoing corticosteroid use (except for subjects who are on stable doses of < 20 mg of prednisone daily [or equivalent] or who are taking corticosteroids for reasons other than cancer)
* Other malignancies (except for adequately treated carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, or basal or squamous cell skin cancer)
* Serious systemic disease, including active infection, uncontrolled hypertension (diastolic blood pressure > 100 mmHg on two consecutive occasions), unstable angina, congestive heart failure, or myocardial infarction or unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia [i.e., atrial fibrillation], paroxysmal supraventricular tachycardia, or controlled hypertension are eligible)
* Liver disease (including viral or other hepatitis), current alcohol abuse, or cirrhosis
* Known human immunodeficiency virus infection
* Pregnancy or lactation
* Major surgery or significant traumatic injury within 3 weeks prior to Day 1
* Inability to comply with study and follow-up procedures
* Any diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the continued use of an investigational drug or that may render the subject at high risk from treatment complications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mika Derynck, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pertuzumab
Started | 3
Completed | 0
Not Completed | 3
Not completed — disease progression | 3

BASELINE CHARACTERISTICS:
Population: Safety population: Participants who received at least 1 dose of pertuzumab.
Arm/Group | Pertuzumab
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event
Time Frame: Baseline to the end of the study (up to 2 years, 5 months)
Population: Safety population: Participants who received at least 1 dose of pertuzumab. Percentage of participants
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab
Number analyzed (Participants) | 3
percentage of participants | 33.3

2. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD)
Description: A best overall response could occur at any time during the study and was determined by Response Evaluation Criteria in Solid Tumors (RECIST). A CR was defined as the disappearance of all target lesions (TL) or the disappearance of all non-TLs and normalization of tumor marker level. A PR was defined as at least a 30% decrease in the sum of the longest diameter (SLD) of TLs, taking as reference the baseline SLD. SD was defined as neither sufficient shrinkage to qualify for a PR nor sufficient increase to qualify for PD, taking as reference the smallest SLD since the treatment started for TLs and the persistence of 1 or more non-TL(s) and/or the maintenance of tumor marker level above normal limits. PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since the treatment started or the appearance of one or more new lesions or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs.
Time Frame: Baseline to the end of the study (up to 2 years, 5 months)
Population: Safety population: Participants who received at least 1 dose of pertuzumab.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab
Number analyzed (Participants) | 3
percentage of participants
  Complete response | 0.0
  Partial response | 0.0
  Stable disease | 33.3
  Progressive disease | 33.3
  Unknown | 33.3

ADVERSE EVENTS:
Description: Safety population: Participants who received at least 1 dose of pertuzumab.
Arm/Group | Pertuzumab
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab (N=3)
EJECTION FRACTION DECREASED (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.